CLINICAL TRIAL: NCT00001883
Title: Quality Control of P-CCMB Cardiopulmonary Exercise Equipment
Brief Title: Quality Control of Cardiopulmonary Exercise Equipment
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990067; 99-H-0067
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2002-10

CONDITIONS: Healthy
Keywords: Treadmill; Bicycle; Lung Function; Physiology; Quality Control; Normal Volunteers

SUMMARY:
This study is designed to make sure exercise equipment used by the National Heart, Lung, and Blood Institute is working properly. Healthy volunteers will be requested to use P-CCMB cardiopulmonary exercise equipment (treadmills and exercise bicycles) two times a month to ensure the machines are functioning properly.

DETAILED DESCRIPTION:
Proper functioning of recently acquired P-CCMB cardiopulmonary exercise equipment will be verified by testing healthy volunteers. In addition, quality control will be verified by performing monthly testing of healthy volunteers as biologic standards.

ELIGIBILITY:
INCLUSION:

Healthy research volunteers who are between 21 and 65 years.

EXCLUSION:

Patients with a history of ischemic or valvular heart disease.

Patients with history of chronic pulmonary disease.

Pregnant women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-03; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sue DY, Wasserman K. Impact of integrative cardiopulmonary exercise testing on clinical decision making. Chest. 1991 Apr;99(4):981-92. doi: 10.1378/chest.99.4.981. No abstract available. PMID 2009806
- [Background] Whipp BJ. The bioenergetic and gas exchange basis of exercise testing. Clin Chest Med. 1994 Jun;15(2):173-92. PMID 8088087
- [Background] Wagner PD. Central and peripheral aspects of oxygen transport and adaptations with exercise. Sports Med. 1991 Mar;11(3):133-42. doi: 10.2165/00007256-199111030-00001. No abstract available. PMID 2047621